CLINICAL TRIAL: NCT00353366
Title: Open, Multicentric, Post-marketing Surveillance Study to Evaluate Safety and Reactogenicity of GSK Bio's Live Attenuated Oral Human Rotavirus (HRV) Vaccine, Rotarix When Administered According to Prescribing Information, in Filipino Subjects Aged at Least 6 Weeks of Age at the Time of First Vaccination
Brief Title: To Evaluate Safety & Reactogenicity of GSK Bio's Human Rotavirus (HRV) Vaccine in Filipino Infants at Least 6 Weeks of Age at First Vaccination
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 103366; 2012-004039-21 (EudraCT Number)
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Results first posted 2011-08-03 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Infections, Rotavirus; Rotavirus Vaccines
Keywords: safety; Post-marketing surveillance (PMS); Rotarix; oral; Filipino; Rotavirus; Gastroenteritis; Human Rotavirus (HRV) vaccine
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — RIX4414 vaccine; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort Group: Subjects received two oral doses of the Rotarix vaccine at the age of 6 weeks
  Interventions: Biological: Rotarix; Other: Data collection

INTERVENTIONS:
Biological: Rotarix — Two doses of the oral vaccine
Other: Data collection — Safety evaluation: recording of adverse events by using diary cards and by non-leading questioning.

SUMMARY:
GSK has submitted a registration file for its live attenuated oral human rotavirus (HRV) vaccine in several countries. In view of its registration in the Philippines, the present study will collect data on the safety of the vaccine in the local target population as per the Bureau of Food and Drugs Directive.

DETAILED DESCRIPTION:
The protocol was amended to reflect a change in the prescribing information. The age of the infants was changed from 6 - 14 weeks to at least 6 weeks at the time of the first vaccination. This protocol posting has been amended in order to comply with FDA AA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits) should be enrolled in the study.
* A Filipino male or female aged at least 6 weeks at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.

Exclusion Criteria:

* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any history of chronic gastrointestinal disease including any uncorrected congenital malformation of the GI tract.
* Any contraindications as stated in the Prescribing Information.

Ages: 6 Weeks to 24 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Filipino subjects aged at least 6 weeks at the time of first vaccination
Sampling Method: Non-Probability Sample
Enrollment: 1439 (Actual)
Dates: Start 2006-11-16 (Actual); Primary Completion 2010-03-31 (Actual); Study Completion 2010-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Philippines (15):
  - GSK Investigational Site, Alabang, Muntinlupa City
  - GSK Investigational Site, Binangonan, Rizal
  - GSK Investigational Site, Cainta, Rizal
  - GSK Investigational Site, City of Muntinlupa
  - GSK Investigational Site, Gen. Trias, Cavite
  - GSK Investigational Site, Imus, Cavite
  - GSK Investigational Site, Los Banos, Laguna
  - GSK Investigational Site, Makati City
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Maybunga, Pasig City
  - GSK Investigational Site, Pasay
  - GSK Investigational Site, Pasig City, Metro Manila
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, Talaba IV, Bacoor, Cavite
  - GSK Investigational Site, Taytay, Rizal

REFERENCES:
- [Background] Bravo L, Chitraka A, Liu A, Choudhury J, Kumar K, Berezo L, Cimafranca L, Chatterjee P, Garg P, Siriwardene P, Bernardo R, Mehta S, Balasubramanian S, Karkada N, Htay Han H. Reactogenicity and safety of the human rotavirus vaccine, Rotarix in The Philippines, Sri Lanka, and India: a post-marketing surveillance study. Hum Vaccin Immunother. 2014;10(8):2276-83. doi: 10.4161/hv.29280. PMID 25424932

RESULTS

PARTICIPANT FLOW:
Groups:
- Rotarix Group: Subjects received 2 doses of Rotarix administered at an interval of not less than 4 weeks between the doses. The first dose was administered at the age of 6 weeks and the vaccination course completed by the age of 24 weeks.
Period: Overall Study
Arm/Group | Rotarix Group
Started | 1439
Completed | 1296
Not Completed | 143
Not completed — Adverse Event | 8
Not completed — Protocol Violation | 12
Not completed — Withdrawal by Subject | 12
Not completed — Lost to Follow-up | 92
Not completed — Other | 19

BASELINE CHARACTERISTICS:
Arm/Group | Rotarix Group
Number analyzed (Participants) | 1439
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 11.2 (3.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 692
  Male | 747

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Grade 2 or 3 Symptoms (Fever, Vomiting or Diarrhea).
Description: Grade 2 or 3 symptoms assessed include fever, vomiting and diarrhea. Grade 2 fever was defined as axillary temperature above 38.0 degrees Celsius (°C) and below or equal to 39.0°C or rectal temperature above 38.5°C and below or equal to 39.5°C. Grade 3 fever was defined as axillary temperature above 39.0°C. Grade 2 vomiting was defined as 2 episodes of vomiting per day. Grade 3 vomiting was defined as at least 3 episodes of vomiting per day. Grade 2 diarrhea was defined as 4-5 looser than normal stools per day. Grade 3 diarrhea was defined as at least 6 looser than normal stools per day.
Time Frame: During the 15-day (Days 0-14) solicited follow-up period after each vaccine dose (Dose 1 and Dose 2).
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects with at least one dose of the Rotarix vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 1439
Subjects
  Grade 2/3;Dose 1 | 147
  Grade 2/3; Dose 2: number analyzed (Participants) | 1304
  Grade 2/3; Dose 2 | 98
  Grade 2/3; Across Doses | 212

2. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited symptoms assessed included cough, diarrhea, fever, irritability, loss of appetite and vomiting. Any = Any reports of the specified symptom irrespective of intensity grade and relationship to vaccination. Grade 3 symptom: symptom that prevented normal activity. Grade 3 loss of appetite = not eating at all, grade 3 fever = axillary temperature > 39.0°C, grade 3 vomiting = ≥ 3 episodes of vomiting/day and grade 3 diarrhea = ≥ 6 looser than normal stools/day. Related = symptom assessed by the investigator as causally related to the vaccination regardless of intensity grade.
Time Frame: During the 15-day solicited follow-up period (Day 0 to Day 14) after each vaccine dose (Dose 1 and Dose 2).
Population: The analysis was performed on the Total Vaccinated cohort , which included all vaccinated subjects with at least one dose of the Rotarix vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 1439
Subjects
  Any Cough; Dose 1 | 311
  Grade 3 Cough; Dose 1 | 13
  Related Cough; Dose 1 | 15
  Any Diarrhea; Dose 1 | 69
  Grade 3 Diarrhea; Dose 1 | 13
  Related Diarrhea; Dose 1 | 26
  Any Temperature; Dose 1 | 130
  Grade 3 Temperature; Dose 1 | 3
  Related Temperature; Dose 1 | 26
  Any Irritability; Dose 1 | 464
  Grade 3 Irritability; Dose 1 | 36
  Related Irritability; Dose 1 | 100
  Any Loss of appetite; Dose 1 | 269
  Grade 3 Loss of appetite; Dose 1 | 4
  Related Loss of appetite; Dose 1 | 74
  Any Vomiting; Dose 1 | 190
  Grade 3 Vomiting; Dose 1 | 44
  Related Vomiting; Dose 1 | 38
  Any Cough; Dose 2 | 256
  Grade 3 Cough; Dose 2: number analyzed (Participants) | 1304
  Grade 3 Cough; Dose 2 | 7
  Related Cough; Dose 2: number analyzed (Participants) | 1304
  Related Cough; Dose 2 | 27
  Any Diarrhea; Dose 2: number analyzed (Participants) | 1304
  Any Diarrhea; Dose 2 | 38
  Grade 3 Diarrhea; Dose 2: number analyzed (Participants) | 1304
  Grade 3 Diarrhea; Dose 2 | 5
  Related Diarrhea; Dose 2: number analyzed (Participants) | 1304
  Related Diarrhea; Dose 2 | 14
  Any Temperature; Dose 2: number analyzed (Participants) | 1304
  Any Temperature; Dose 2 | 130
  Grade 3 Temperature; Dose 2: number analyzed (Participants) | 1304
  Grade 3 Temperature; Dose 2 | 4
  Related Temperature; Dose 2: number analyzed (Participants) | 1304
  Related Temperature; Dose 2 | 24
  Any Irritability; Dose 2: number analyzed (Participants) | 1304
  Any Irritability; Dose 2 | 307
  Grade 3 Irritability; Dose 2: number analyzed (Participants) | 1304
  Grade 3 Irritability; Dose 2 | 24
  Related Irritability; Dose 2: number analyzed (Participants) | 1304
  Related Irritability; Dose 2 | 71
  Any Loss of appetite; Dose 2: number analyzed (Participants) | 1304
  Any Loss of appetite; Dose 2 | 193
  Grade 3 Loss of appetite; Dose 2: number analyzed (Participants) | 1304
  Grade 3 Loss of appetite; Dose 2 | 5
  Related Loss of appetite; Dose 2: number analyzed (Participants) | 1304
  Related Loss of appetite; Dose 2 | 43
  Any Vomiting; Dose 2: number analyzed (Participants) | 1304
  Any Vomiting; Dose 2 | 113
  Grade 3 Vomiting; Dose 2: number analyzed (Participants) | 1304
  Grade 3 Vomiting; Dose 2 | 13
  Related Vomiting; Dose 2: number analyzed (Participants) | 1304
  Related Vomiting; Dose 2 | 22
  Any Cough; Across Doses | 443
  Grade 3 Cough; Across Doses | 18
  Related Cough; Across Doses | 39
  Any Diarrhea; Across Doses | 93
  Grade 3 Diarrhea; Across Doses | 18
  Related Diarrhea; Across Doses | 36
  Any Temperature; Across Doses | 226
  Grade 3 Temperature; Across Doses | 7
  Related Temperature; Across Doses | 48
  Any Irritability; Across Doses | 545
  Grade 3 Irritability; Across Doses | 51
  Related Irritability; Across Doses | 130
  Any Loss of appetite; Across Doses | 351
  Grade 3 Loss of appetite; Across Doses | 8
  Related Loss of appetite; Across Doses | 93
  Any Vomiting; Across Doses | 240
  Grade 3 Vomiting; Across Doses | 54
  Related Vomiting; Across Doses | 49

3. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any was defined as an adverse event (AE) reported in addition to those solicited during the clinical study. Any solicited symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: During the 31-day follow-up period (Day 0 to Day 30) after any vaccine dose.
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one dose of the Rotarix vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 1439
Subjects | 352

4. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: Serious adverse events (SAEs) assessed include medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the study period (Day 0 to one month post-Dose 2).
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Rotarix Group
Number analyzed (Participants) | 1439
Participants | 33

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: during the entire study period; Solicited local and general symptoms: During the 15-day (Days 0-14) post-vaccination period; Unsolicited symptoms: During the 31-day (Days 0-30) post-vaccination period.
Arm/Group | Rotarix Group
All-Cause Mortality (participants affected / at risk) | 0/1439
Serious Adverse Events (participants affected / at risk) | 33/1439
Other Adverse Events (participants affected / at risk) | 827/1439
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=1439)
Bronchopneumonia (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 5
Amoebic dysentery (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Amoebiasis (Infections and infestations) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea infections (Infections and infestations) | 1
Exanthema subitum (Skin and subcutaneous tissue disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Hypersomnia (Nervous system disorders) | 1
Hypophagia (Nervous system disorders) | 1
Intussusception (Gastrointestinal disorders) | 1
Milk anyergy (Immune system disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia bacterial (Infections and infestations) | 1
Roseola (Infections and infestations) | 1
Urinary tract infection enterococcal (Infections and infestations) | 1
Viral rash (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=1439)
Cough (General disorders) | 443
Diarrhea (Gastrointestinal disorders) | 93
Fever (General disorders) | 226
Irritability (General disorders) | 545
Loss of appetite (General disorders) | 351
Vomiting (General disorders) | 240

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.